CLINICAL TRIAL: NCT02870842
Title: Effects of Fraction of Inspired Oxygen on Atelectasis in Mechanically Ventilated Children
Brief Title: Fraction of Inspired Oxygen and Atelectasis in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-1607-150-778
Record Dates: First submitted 2016-08-14; First posted 2016-08-17 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Atelectasis
Keywords: ultrasonography; child; perioperative period; general anesthesia; lung
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Perform recruitment maneuver with fraction of inspired oxygen (FiO2) of 1.0 after intubation under lung ultrasound guidance and maintain FiO2 of 0.6 during the general anesthesia.
  Interventions: Device: Lung ultrasound; Other: Respiratory management
- Low FiO2 (Active Comparator): Perform recruitment maneuver with low FiO2 of 0.3 after intubation under lung ultrasound guidance and maintain FiO2 of 0.3 during the general anesthesia.
  Interventions: Device: Lung ultrasound; Other: Respiratory management

INTERVENTIONS:
Device: Lung ultrasound — Lung ultrasound on both hemithorax in supine position
Other: Respiratory management — Appropriate respiratory managements depending on the lung ultrasound findings

SUMMARY:
Investigators hypothesized that maintaining low fraction of inspired oxygen would be beneficial to prevent anesthesia-induced atelectasis in mechanically ventilated children undergoing general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Expected operation time between 1 to 3 hours under general anesthesia
* Mechanically ventilated after endotracheal intubation

Exclusion Criteria:

* Cardiac, thoracic, abdominal surgery
* History of surgery on the lungs
* Laparoscopic surgery
* Abnormal preoperative chest radiograph findings including atelectasis, pneumothorax, pleural effusion, and pneumonia
* Considered inappropriate by the investigator

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2016-09; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative atelectasis | within the first day after the surgery

SECONDARY OUTCOMES:
Incidence of atelectasis after endotracheal intubation | from the moment of endotracheal intubation until the end of surgery, up to 4 hours
Intraoperative incidence of pulse oximetry (SpO2) ≤ 95% (or 10% below the baseline value) | from the induction of general anesthesia until the end of the surgery, up to 4 hours
Postoperative incidence of pulse oximetry (SpO2) ≤ 95% (or 10% below the baseline value) | within the first day after the surgery
Postoperative incidence of fever (≥37.5℃) | within the first day after the surgery
Postoperative incidence of respiratory complications | within the first day after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Acosta CM, Maidana GA, Jacovitti D, Belaunzaran A, Cereceda S, Rae E, Molina A, Gonorazky S, Bohm SH, Tusman G. Accuracy of transthoracic lung ultrasound for diagnosing anesthesia-induced atelectasis in children. Anesthesiology. 2014 Jun;120(6):1370-9. doi: 10.1097/ALN.0000000000000231. PMID 24662376
- [Background] Edmark L, Auner U, Enlund M, Ostberg E, Hedenstierna G. Oxygen concentration and characteristics of progressive atelectasis formation during anaesthesia. Acta Anaesthesiol Scand. 2011 Jan;55(1):75-81. doi: 10.1111/j.1399-6576.2010.02334.x. Epub 2010 Oct 29. PMID 21039356
- [Background] Akca O, Podolsky A, Eisenhuber E, Panzer O, Hetz H, Lampl K, Lackner FX, Wittmann K, Grabenwoeger F, Kurz A, Schultz AM, Negishi C, Sessler DI. Comparable postoperative pulmonary atelectasis in patients given 30% or 80% oxygen during and 2 hours after colon resection. Anesthesiology. 1999 Oct;91(4):991-8. doi: 10.1097/00000542-199910000-00019. PMID 10519502
- [Background] Martin JB, Garbee D, Bonanno L. Effectiveness of positive end-expiratory pressure, decreased fraction of inspired oxygen and vital capacity recruitment maneuver in the prevention of pulmonary atelectasis in patients undergoing general anesthesia: a systematic review. JBI Database System Rev Implement Rep. 2015 Sep 16;13(8):211-49. doi: 10.11124/jbisrir-2015-1410. PMID 26455945